CLINICAL TRIAL: NCT01377012
Title: A Randomized, Double-blind, Placebo-controlled Study of Secukinumab to Demonstrate the Efficacy at 24 Weeks and to Assess the Safety, Tolerability and Long Term Efficacy up to 2 Years in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Anti-TNFα Agents (CAIN457F2302) and a Three Year Extension Study to Evaluate the Long Term Efficacy, Safety and Tolerability of Secukinumab in Patients With Active Rheumatoid Arthritis (CAIN457F2302E1)
Brief Title: Efficacy at 24 Weeks and Safety, Tolerability and Long Term Efficacy up to 2 Years of Secukinumab (AIN457) in Patients With Active Rheumatoid Arthritis and an Inadequate Response to Anti-TNFα Agents
Acronym: REASSURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2302/E1; 2011-000275-13 (EudraCT Number); NCT01901900 (obsolete NCT alias)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; ACR; inflammatory joints
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AIN457 10mg/kg-75mg (Experimental): Participants received AIN457 i.v. (10 mg/kg) at Baseline (BSL), Weeks 2 and 4 then AIN457 75 mg s.c. at Week 8 and injected every 4 weeks
  Interventions: Biological: Secukinumab (AIN457)
- AIN457 10mg/kg-150mg (Experimental): Participants received AIN457 i.v. (10 mg/kg) at BSL, Weeks 2 and 4 then AIN457 150 mg s.c. at Week 8 and injected every 4 weeks
  Interventions: Biological: Secukinumab (AIN457)
- Placebo (Placebo Comparator): Participants received matching placebo to AIN457 until week 16 or week 24 based on responder status (>= 20% reduction in tender and swollen joint count). Non-responders were switched to active treatment at week 16. Responders were switched to active treatment at week 24
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab (AIN457) — AIN457 (Secukinumab) is a human monoclonal antibody. Secukinumab binds and reduces the activity of Interleukin 17 (IL- 17). AIN457 was given as i.v. (10mg/kg) at baseline, week 2 and week 4, and then s.c. (75 or 150mg) every 4 weeks starting at week 8.
  Other Names: AIN457
  Arms: AIN457 10mg/kg-150mg; AIN457 10mg/kg-75mg
Biological: Placebo — Placebo was given as i.v. at baseline, week 2 and week 4, and then s.c. every 4 weeks starting at week 8.
  Arms: Placebo

SUMMARY:
The core and extension studies assessed the safety and efficacy of secukinumab when added to a background therapy in patients with active rheumatoid arthritis who are intolerant to or have had an inadequate response to anti-TNF-α agents. Patients received either secukinumab, placebo. The core study was completed. However, the extension study was terminated early (unrelated to safety) due to the results of study AIN457F2309, which indicated the efficacy of AIN457 was not comparable to the currently available RA treatment, abatacept, thus leading to closing of the AIN457 RA program.

DETAILED DESCRIPTION:
CAIN457F2302 (Core Study): Completed Sep 9 2015

CAIN457F2302E1 (Extension study): terminated early May 26 2015, ((unrelated to safety) due to the results of study AIN457F2309, which indicated the efficacy of AIN457 was not comparable to the currently available RA treatment, abatacept, thus leading to closing of the AIN457 RA program.

ELIGIBILITY:
Inclusion criteria:

* Male or non-pregnant, non-lactating female patients
* Presence of RA classified by American College of Rheumatology (ACR) 2010 revised criteria for at least 3 months before screening
* At Baseline: Disease activity criteria defined by ≥ 6 tender joints out of 68 and ≥6 swollen joints out of 66 with at least 1 of the following at screening:
* Anti-Cyclic Citrullinated Peptide (CCP) antibodies positive OR

Rheumatoid Factor positive and with at least 1 of the following at screening:

* High sensitivity C-reactive protein (hsCRP) ≥ 10 mg/L OR Erythrocyte sedimentation rate (ESR) ≥ 28 mm/1st hr
* Patients must have been taking at least one anti-TNF-α agent given at an approved dose for at least 3 months before randomization and have experienced an inadequate response to treatment or have been intolerant to at least one administration of an anti-TNF-α agent
* Patients must be taking MTX for at least 3 months before randomization and have to be on a stable dose at least 4 weeks before randomization (7.5 to 25 mg/week For Japan only: 6 to 25 mg/week)

Exclusion criteria:

* Chest x-ray with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician RA patients functional status class IV according to the ACR 1991 revised criteria
* Patients who have ever received biologic immunomodulating agents except for those targeting TNFα
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20, investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19)
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (127):
- United States (37):
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Paradise Valley, Arizona
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Canton, Georgia
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Eagan, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Gallipolis, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
- Argentina (8):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires F.D.
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
- Canada (3):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, St. Catharines, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Colombia (3):
  - Novartis Investigative Site, Bucaramanga, Colombia
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Veszprém
- India (9):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Amravati, Maharashtra
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ajmer, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Secunderabad, Telangana
- Italy (5):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pieve di Coriano, MN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
- Japan (35):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Yotsukaidō, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Takasaki, Gunma
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Taihaku-ku, Miyagi
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Tsukubo-gun, Okayama-ken
  - Novartis Investigative Site, Hannan, Osaka
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Fuji, Shizuoka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
- Mexico (4):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Culiacán, Sinaloa
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Puerto Rico (2):
  - Novartis Investigative Site, Ponce
  - Novartis Investigative Site, San Juan
- Thailand (6):
  - Novartis Investigative Site, Bangkok, Bangkok
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Songkhla
- Novartis Investigative Site, Ankara, Turkey, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Salisbury

REFERENCES:
- [Derived] Huang Y, Fan Y, Liu Y, Xie W, Zhang Z. Efficacy and safety of secukinumab in active rheumatoid arthritis with an inadequate response to tumor necrosis factor inhibitors: a meta-analysis of phase III randomized controlled trials. Clin Rheumatol. 2019 Oct;38(10):2765-2776. doi: 10.1007/s10067-019-04595-1. Epub 2019 May 14. PMID 31087226
- [Derived] Tahir H, Deodhar A, Genovese M, Takeuchi T, Aelion J, Van den Bosch F, Haemmerle S, Richards HB. Secukinumab in Active Rheumatoid Arthritis after Anti-TNFalpha Therapy: A Randomized, Double-Blind Placebo-Controlled Phase 3 Study. Rheumatol Ther. 2017 Dec;4(2):475-488. doi: 10.1007/s40744-017-0086-y. Epub 2017 Nov 14. PMID 29138986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At baseline, participants were randomized to 1 of 3 treatment groups. Placebo non- responders at week 16 were re-randomized to receive AIN457 75mg or AIN457 150mg. Placebo responders at Week16 were re-randomized to receive AIN457 75mg or AIN457 150mg at Week 24.
Groups:
- AIN457 10mg/Kg-75mg: Participants received AIN457 i.v. (10 mg/kg) at Baseline (BSL), Weeks 2 and 4 then AIN457 75 mg s.c. at Week 8 and injected every 4 weeks up to Week 100, then AIN457 150 mg s.c. starting at week 104
Period: Core Study
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Started | 210 | 213 | 214
wk16 Re-randomized to AIN 75mg NR | 0 | 0 | 56 (NR=Non-responder)
wk16 Re-randomized to AIN 150mg NR | 0 | 0 | 53
wk 24 Re-randomized to AIN 75 mg Res | 0 | 0 | 38 (Res= responder)
wk 24 Re-randomized to AIN 150 mg Res | 0 | 0 | 34
Completed | 76 | 81 | 80
Not Completed | 134 | 132 | 134
Not completed — Study terminated by Sponsor | 47 | 54 | 46
Not completed — Technical problems | 1 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 23 | 18
Not completed — Protocol Violation | 7 | 3 | 2
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Physician Decision | 5 | 4 | 10
Not completed — Non-Compliant with study treatment | 0 | 0 | 1
Not completed — No Longer require treatment | 0 | 0 | 1
Not completed — Lost to Follow-up | 7 | 5 | 4
Not completed — Lack of Efficacy | 41 | 28 | 37
Not completed — Death | 1 | 1 | 1
Not completed — Adverse Event | 10 | 14 | 13
Period: Extension Study, Weeks 104-260
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Started | 57 | 71 | 68
Completed | 0 | 0 | 0
Not Completed | 57 | 71 | 68
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Study terminated by sponsor | 52 | 69 | 63
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo | Total
Number analyzed (Participants) | 210 | 213 | 214 | 637
Age, Customized [Number; unit: Particpants]
  <65 years | 177 | 176 | 182 | 535
  >=65 years | 33 | 37 | 32 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 188 | 182 | 556
  Male | 24 | 25 | 32 | 81

OUTCOME MEASURES:

1. Secondary Outcome: Core Study: Change From Baseline and Week 24 in Stanford Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: Participants from the full analysis set were considered for the analysis. Participants with measurements at both baseline and week 24 were analyzed. The full analysis set was comprised of all randomized participants (excluding mis-randomized participants) who were assigned to study treatment.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 171 | 188 | 71
Score on a scale | -0.35 (0.039) | -0.35 (0.038) | -0.24 (0.051)

2. Secondary Outcome: Core Study: Change From Baseline at Week 24 in Van Der Heijde Total Modified Sharp Score
Description: Separate radiographs of each hand/wrist and each foot were taken at basline and Week 24. The radiographs were assessed using the van der Heijde modified Sharp score. The change in the Van der Heijde modified Sharp score is calculated against the baseline value. The total van der Heide modified Sharp score goes from 0 to 448, the bigger the change, the worse it is for the patient.
Time Frame: Week 24
Population: Participants from the full analysis set were considered for the analysis. Participants with measurements at both baseline and week 24 were analyzed.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 60 | 67 | 83
Score on a scale | 0.59 (0.62) | 0.83 (0.68) | 1.73 (0)

3. Secondary Outcome: Core Study Percentage of Patients Achieving Major Clinical Response (Continuous Six-month Period of ACR70 Response During the 1 Year Period) at Week 52
Description: The major clinical response is defined as continuous six-month period of ACR70 response during the 1 year period. ACR70 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 70% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). The ACR70 response results at week 24 used non-responder imputation.
Time Frame: 52 week
Population: The Full analysis set (FAS) comprised all patients who were randomized and to whom study treatment had been assigned. N=The total number of subjects in the treatment groups with evaluation
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 210 | 213 | 214
Percentage of Participants | 2.4 | 0.9 | 1.4

4. Primary Outcome: Core Study: Percentage of Participants Achieving an American College of Rheumatology Response 20 (ACR20) at Week 24
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). The ACR20 response results at week 24 used non-responder imputation.
Time Frame: Week 24
Population: The Full analysis set (FAS) comprised all patients who were randomized and to whom study treatment had been assigned.
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 210 | 213 | 214
Percentage of Participants | 35.2 | 35.2 | 19.6
Statistical Analysis 1: Comparison: AIN457 10mg/Kg-75mg vs Placebo; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.4 to 3.4]
Statistical Analysis 2: Comparison: AIN457 10mg/Kg-150mg vs Placebo; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.4 to 3.4]

5. Secondary Outcome: Extension Phase: Change in Baseline of RA Disease Activity as Measured by Disease Activity Score (DAS28)
Description: The DAS28 score is a measure of RA disease activity calculated using variables such as swollen joint count, the Erythrocyte Sedimentation Rate (ESR) and patient reported assessment of health.
  Using this data, the DAS28 calculation provides a number on a scale from 0-10 indicating the current activity of a patient's RA. A DAS28 score above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 score lower than 2.6.
Time Frame: week 260
Population: The outcome measures were not analyzed, as a result of the lack of efficacy found in study AIN457F2309 and as per changes to the planned analysis plan for CAIN457f2302/E1
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Extension Phase: Proportion of Subjects Achieving Low Disease Activity and Good/Moderate European League Against Rheumatism (EULAR) Responses
Description: Low Disease Activity is defined as DAS28 ≤ 3.2. EULAR good response requires an improvement of > 1.2 in the DAS28 score with a present score of ≤3.2; EULAR moderate response is defined as an improvement of >0.6 to ≤1.2 in DAS28 and a present score of ≤5.1; or an improvement of >1.2 and a present score of >3.2.
Time Frame: up to week 260
Population: as for outcome 5
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Extension Phase: Proportion of Subjects Achieving ACR/(EULAR) Remission
Description: ACR/EULAR remission is defined as SDAI ≤ 3.3, where SDAI is a measure of disease activity in RA based on 28 tender and swollen joint counts, CRP, Physician and Patient's Global Assessments of Disease
Time Frame: up to week 260
Population: as for outcome 5
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Extension Phase: Changes in Baseline of Quality of Life (Qol) Outcomes Measured by Medical Outcome Short Form SF-36 v2
Description: Short Form Health Survey (SF-36) consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed.
Time Frame: Baseline, up to week 260
Population: as for outcome 5
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Extension Phase: Immunogenicity Against Secukinumab
Time Frame: up to week 260
Population: as for outcome 5
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Extension Phase: Percentage of Patients Achieving a American College of Rheumatology Response ACR20, ACR50 and ACR70
Time Frame: up to week 260
Population: as for outcome 5
Arm/Group | AIN457 10mg/Kg-75mg | AIN457 10mg/Kg-150mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety data is reported (core + extension). Events of placebo patients post switch to active were counted in active group. The "any AIN457 75 mg" "any AIN457 150 mg" groups have all patients originally randomized to group and all placebo patients re-randomized to group, respectively. The "any AIN457 150 mg" group contains all extension patients.
Groups:
- Any AIN457 75 mg: Group contains all patients who received AIN 75mg during core period of the study. Includes : participants who were randomized to receive AIN457 i.v (10 mg/kg) at Baseline (BSL), Weeks 2 and 4 then AIN457 75 mg s.c. at Week 8 injected every 4 weeks + participants who were re-randomized to switch from placebo to AIN457 75 mg at week 16 or week 24 of core study
- Any AIN457 150 mg: Group contains all patients from the core and the extension that ever received AIN 150mg. This includes : participants who were randomized to AIN457 150 mg arm to receive AIN457 i.v. (10 mg/kg) at BSL, Weeks 2 and 4 then AIN457 150 mg s.c. at Week 8 injected every 4 weeks + participants who were re-randomized to switch from placebo to AIN457 150 mg at week 16 or week 24 + participants who completed core study in any arm and continued in the extension study to receive AIN457 150 mg as open-label study drug
- Placebo: Participants received matching placebo to AIN457 until week 16 or week 24 based on responder status (>= 20% reduction in tender and swollen joint count). Non-responders were switched to active treatment at week 16 of core. Responders were switched to active treatment in week 24 of core
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 33/301 | 48/392 | 9/214
Other Adverse Events (participants affected / at risk) | 184/301 | 225/392 | 91/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=301) | Any AIN457 150 mg (N=392) | Placebo (N=214)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1
Sudden death (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 5 | 0
Gangrene (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Joint tuberculosis (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 2
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 3 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Occult blood positive (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Carotid artery insufficiency (Nervous system disorders) | 1 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Cerebellar embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=301) | Any AIN457 150 mg (N=392) | Placebo (N=214)
Anaemia (Blood and lymphatic system disorders) | 9 | 11 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 8 | 2
Constipation (Gastrointestinal disorders) | 6 | 13 | 5
Dental caries (Gastrointestinal disorders) | 4 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 22 | 6
Nausea (Gastrointestinal disorders) | 6 | 15 | 6
Stomatitis (Gastrointestinal disorders) | 6 | 8 | 1
Vomiting (Gastrointestinal disorders) | 4 | 8 | 5
Oedema peripheral (General disorders) | 7 | 8 | 1
Pyrexia (General disorders) | 8 | 13 | 4
Bronchitis (Infections and infestations) | 15 | 31 | 1
Conjunctivitis (Infections and infestations) | 4 | 8 | 0
Cystitis (Infections and infestations) | 4 | 15 | 0
Gastroenteritis (Infections and infestations) | 4 | 13 | 2
Herpes zoster (Infections and infestations) | 8 | 9 | 1
Influenza (Infections and infestations) | 11 | 10 | 2
Nasopharyngitis (Infections and infestations) | 49 | 63 | 14
Pharyngitis (Infections and infestations) | 23 | 18 | 5
Sinusitis (Infections and infestations) | 6 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 25 | 39 | 10
Urinary tract infection (Infections and infestations) | 28 | 33 | 8
Contusion (Injury, poisoning and procedural complications) | 5 | 10 | 2
Alanine aminotransferase increased (Investigations) | 7 | 10 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 9 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 16 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 11 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 9 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 20 | 17 | 11
Dizziness (Nervous system disorders) | 6 | 8 | 3
Headache (Nervous system disorders) | 14 | 18 | 10
Insomnia (Psychiatric disorders) | 3 | 12 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 18 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 8 | 3
Hypertension (Vascular disorders) | 18 | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.